CLINICAL TRIAL: NCT01079611
Title: Non-invasive Assessments of Central Venous Pressure by Ultrasound and Clinical Examination: a Prospective Comparative Study
Brief Title: Non-invasive Assessments of Central Venous Pressure
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Heiko Uthoff, Principal Investigator, University Hospital, Basel, Switzerland
Other Study IDs: CVP1
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Venous Pressure, Central; Ultrasonic Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Estimates of central venous pressure (CVP) can be very helpful in guiding fluid therapy in the intensive care unit, operating room or emergency room. Current standard technique for CVP assessment is invasive, requiring insertion of a catheter into a subclavian, internal jugular or peripheral vein. Several ultrasound based and clinical methods have been described as potential non-invasive alternatives to assess CVP.

Aim: To prospectively evaluate the accuracy of CVP assessment by a) inferior vena cava diameter and collapsibility b) internal jugular vein diameter c) compression sonography of a forearm vein and d) clinical assessment of peripheral vein collapse in comparison to invasive CVP measurement.

Study design: single center, prospective observational study

Patients and Methods:

We will examine 77 consecutive patients with invasive venous access and invasive hemodynamic monitoring at the surgical intensive care unit (ICU). After obtaining informed consent, ultrasound examinations of the inferior vena cava, internal jugular vein and compression sonography of a forearm vein as well as clinical evaluation of peripheral vein collapsibility will be performed in a random sequence by different experienced examiner. Invasive CVP is recorded simultaneously to each measurement. Examiners are blinded to clinical parameters and results of previous CVP measurements.

Primary endpoint: Accuracy of each non-invasive method to determine CVP defined by invasively measured CVP.

Secondary endpoint: Comparison of the feasibility of each non-invasive method.

Expected results: We hypothesize that sonographic measurement of inferior vena cava diameter, internal jugular vein diameter and compression sonography of a forearm vein as well as clinical assessment of peripheral vein collapsibility are reliable methods for CVP determination in comparison to invasive CVP measurement.

Significance: The validation and comparison of sonographic / clinic CVP assessment would enable clinicians to choose an accurate non-invasive method to assess volume status which is an important adjunct in the management of many critically ill patients. The non-invasiveness of these methods broadens the feasibility to measure CVP and may guide fluid therapy in new patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients age greater than 18 years are study candidates if they need central venous access and invasive hemodynamic monitoring, according to the discretion of the treating physician.
* Informed consent is given.

Exclusion Criteria:

* Patients are ineligible if they have a history of neck or body radiotherapy and/or previous or active upper-extremity deep venous thrombosis.
* Informed consent is not given.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This single center, prospective observational study will be performed at the surgical intensive care unit (ICU) of the tertiary care teaching hospital of the University of Basel. ICU, rather than Emergency Department patients will be consecutively enrolled because of the higher prevalence of CVP catheters and the higher likelihood of clinical stability (by means of hemodynamic parameters, therapeutic interventions etc.).
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Uthoff, M.D., Principal Investigator — University Hospital Basel, Angiology; Kurt A Jaeger, M.D., Principal Investigator — University Hospital Basel, Angiology
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Result] Uthoff H, Siegemund M, Aschwanden M, Hunziker L, Fabbro T, Baumann U, Jaeger KA, Imfeld S, Staub D. Prospective comparison of noninvasive, bedside ultrasound methods for assessing central venous pressure. Ultraschall Med. 2012 Dec;33(7):E256-E262. doi: 10.1055/s-0031-1299506. Epub 2012 Jun 1. PMID 22660962